CLINICAL TRIAL: NCT05940896
Title: Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of Disitamab Vedotin Intravenously Combined With Radiotherapy in the Treatment of Locally Advanced Solid Tumors With HER2 Expression Phase 1 Study
Brief Title: RC48-ADC Combined With Radiotherapy in the Treatment of Locally Advanced Solid Tumors With HER2 Expression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C019
Record Dates: First submitted 2023-05-08; First posted 2023-07-11 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumor
Keywords: HER2 expression; solid tumor
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Intervention Model Description: DV is given intravenously once every 2 weeks, (dose escalation plan: 1.0mg/kg, 1.5mg/kg, 2.0mg/kg, 2.5mg/kg). DV will be administered at least 2 times during the treatment, and the final DV dose needs to be completed before the last radiotherapy.
  Concurrent standard radiotherapy for solid tumors is given for 5-7 weeks, 5 times per week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): DV is given intravenously once every 2 weeks, (dose escalation plan: 1.0mg/kg, 1.5mg/kg, 2.0mg/kg, 2.5mg/kg). DV will be administered at least 2 times during the treatment, and the final DV dose needs to be completed before the last radiotherapy.
  Interventions: Drug: Disitamab vedotin

INTERVENTIONS:
Drug: Disitamab vedotin — Disitamab Vedotin intravenously combined with radiotherapy (concurrent)
  Other Names: RC48-ADC

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of Disitamab Vedotin(DV, RC48-ADC) intravenously combined with radiotherapy in the treatment of locally advanced solid tumors with HER2 expression

DETAILED DESCRIPTION:
This study is a single arm, open, single site clinical study aimed at evaluating the safety, tolerability, pharmacokinetic characteristics, and efficacy of Disitamab Vedotin intravenously combined with radiotherapy in the treatment of locally advanced solid tumors with HER2 expression. Unresectable locally advanced solid tumor patients whose SOC is concurrent chemoradiation but ineligible or refuse to standard chemotherapy should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed informed consent,
2. Male or female, aged ≥18 years,
3. Predicted survival ≥ 12 weeks;
4. Based on the investigator's evaluation (histopathological classification and clinical staging), patients with locally advanced solid tumors (head and neck squamous cell carcinoma, esophageal carcinoma, urothelium carcinoma, cervical carcinoma, etc), whose SOC is concurrent chemoradiation and cannot be surgically removed, are ineligible or refuse the standard chemotherapy.
5. The subject has not been given any anti-tumor systemic therapy or radiotherapy for locally advanced solid tumors in the past
6. HER2 expression is confirmed by the site: IHC 1+, 2+or 3+;
7. At least one measurable lesion according to RECIST 1.1.
8. ECOG performance status score of 0 or 1;
9. Adequate heart, bone marrow, liver, and kidney functions, which should meet the following standards within 7 days before the study drug is given (based on the normal values of the site) :

   Left ventricular ejection fraction ≥ 50%; Hemoglobin ≥ 9g/dL; Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L； Platelets ≥ 100 × 10^9/L； Serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); ALT and AST ≤ 2.5 × ULN； Blood creatinine ≤ 1.5 × ULN or calculate creatinine clearance rate (CrCl) ≥ 50 mL/min according to Cockcroft Fault formula method;
10. Female subjects: should be surgically sterilized, postmenopausal, or agree to use a medically approved contraceptive (such as an intrauterine device, contraceptives, or condoms) during study treatment and within 6 months after the end of study, and their blood pregnancy test must be negative within 7 days prior to study enrollment and they must be non-lactating. Male subjects: should be surgically sterile, or agree to use a medically approved contraceptive during study treatment and within 6 months after the end of study;
11. Willing and able to comply with the schedules of the trial and follow-up procedures.

Exclusion Criteria:

1. Received anti-tumor therapy before this study, including radiotherapy, target therapy, immunotherapy, and any anti-tumor clinical studies;
2. The subject was given a major surgery and did not fully recover within 4 weeks prior to the study;
3. Serum virology examination (based on the normal value of the site):

   HBsAg or HBcAb test results are positive, while HBV DNA copy is detected as positive; The HCVAb test result is positive (only when the PCR test result for HCV RNA is negative, can it be selected for this study); The HIVAb test result is positive.
4. The subject was given live vaccine within 4 weeks before the study drug is given or planed to receive any vaccine during the study period (except for Covid-19 vaccine);
5. Heart failure≥ 3 grade（NYHA）
6. Serious arteriovenous thrombotic events or cardiovascular and cerebrovascular accidents, such as deep vein thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc., occurred within one year before the study drug is given, except for lacunar cerebral infarction without symptoms or clinical intervention;
7. There are active or progressive infections that require systematic treatment, such as active pulmonary tuberculosis;
8. There are systemic diseases that have not been controlled stably as judged by the investigator, including diabetes, hypertension, cirrhosis, interstitial pneumonia, obstructive pulmonary disease, etc;
9. Active autoimmune diseases that require systematic treatment (such as the use of immunomodulators, corticosteroids, or immunosuppressants) prior to the start of drug administration, allowing for related alternative treatments (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for renal or pituitary dysfunction);
10. Patients with other malignant tumors within 5 years prior to the start of study administration;
11. Previously received other antibody conjugated drug treatments;
12. Those who are known to be allergic to recombinant humanized anti HER2-ADC and components;
13. Pregnant or lactating women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
DLT | First DV dose to 28 days after the last RT
  Dose limiting toxicity (DLT)
AE | First DV dose to 90 days after the last RT
  the incidence and severity of adverse events (AE);

SECONDARY OUTCOMES:
PK Characterize | Cycle1Day1 to Cycle1Day8 (each cycle is 14 days)
  The concentration of DV binding antibodies, total antibodies, and free MMAE.
Immunogenicity assessment | Cycle1Day1 to Cycle1Day8 (each cycle is 14 days)
  Anti-RC48 antibodies
ORR | approximately 2 years from the first dose
  (RECIST 1.1 standard, evaluated by investigators): objective response rate (ORR), the relationship between HER2 expression and therapeutic efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer hospital &Institute, Jinan, Shandong, China